CLINICAL TRIAL: NCT05117424
Title: The Impact of Cardiometabolic Factors on Coronary Artery and Cardiovascular Diseases: a Prospective Cohort Study
Brief Title: CArdioMetabolism and Atherosclerotic PlaqUe progreSsion
Acronym: CAMPUS
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, RUIYAN ZHANG, Professor, Ruijin Hospital
Other Study IDs: RJH-CAMPUS
Record Dates: First submitted 2021-10-19; First posted 2021-11-11 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus, Type 2; Dyslipidemias; Obesity; Metabolic Syndrome
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 2; Dyslipidemias; Obesity; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Blood samples to determine apoA-I glycation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Systematic metabolic diseases are closely related to prevalence and progression of atherosclerosis. This prospective cohort consecutively enrolls patients with coronary artery disease compliacted with metabolic abnormalities such as diabtetes, prediabetes, obesity, chronic kidney disease and hyperuricemia.

DETAILED DESCRIPTION:
CArdioMetabolism and Atherosclerotic PlaqUe progreSsion (CAMPUS) study is a single center, prospective cohort study to investigate the impact of cardiometabolic factors on coronary diseases. This study consecutively enrolls patients with coronary artery diseases complicatied with metabolic abnormalities, including diabetes, prediabetes, obesity, chronic kidney disease and hyperuricemia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Established coronary artery disease or metabolic disorders, including:

  1. Type 2 diabetes diagnosed by one of the following criteria:

     HbA1c >/= 6.5% Fasting plasma glucose >/= 7.0 mmol/l (confirmed) 2h plasma glucose value during OGTT >/= 11.1 mmol/l Already receiving glucose-lowering agents
  2. Prediabetes
  3. Obesity
  4. Chronic kidney disease
  5. Hyperuricemia
  6. Dyslipidemia

Exclusion Criteria:

* Severe liver failure (Child-Pugh grade B to C)
* Severe anemia (hemoglobin < 60g/L)
* Familial hypercholesterolemia
* Active malignant tumor
* Active autoimmune diseases on corticosteroids
* Acute or chronic infection
* Life expectancy < 1 year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a single-center cohort study. Patients with metabolic disorders (as listed in eligibility criteria) and suspected coronary artery disease undergone coronary angiography at Ruijin Hospital, Shanghai, China are consecutively enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Coronary plaque progression | 12 months
  Assessed by coronary angiography and QCA
Coronary lesion severity | 12 months
  Assessed by coronary angiography and QCA

SECONDARY OUTCOMES:
Coronary plaque characteristics | 12 months
  Assessed by intravascular imaging (IVUS or OCT)
Cardiovascular events | up to 5 years
  The incidence of MACCE (major adverse cardio and cerebral vascular events), lesion associated events (target lesion myocardial infarction, target lesion faliure, target vessel revascularization, etc.)

OTHER OUTCOMES:
Diabetic complications | up to 5 years
  Prevalence of diabetic complications, including peripheral artery disease, retinopathy, nephropathy, encephalopathy.
Glycated modifications of lipoproteins | up to 2 years
  Glycated modifications of lipoproteins in patients, such as ApoA-I glycation.
Lipoprotein function assessment | up to 2 years
  HDL functions, including reverse cholesterol transport assessed by cholesterol efflux capacity, anti-inflammatory function, and anti-oxidation function

CONTACTS AND LOCATIONS:
Overall Officials: Lin Lu, M.D., Ph.D., Study Director — Ruijin Hospital, Shanghai Jiaotong School of Medicine; Fenghua Ding, M.D., Ph.D., Study Chair — Ruijin Hospital, Shanghai Jiaotong School of Medicine; Ruiyan Zhang, M.D., Ph.D., Principal Investigator — Ruijin Hospital, Shanghai Jiaotong School of Medicine
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China